CLINICAL TRIAL: NCT00308269
Title: Protocol EC-FV-01: A Phase 1 Study of EC145 Administered in Weeks 1 and 3 of a 4-Week Cycle
Brief Title: Study of Vintafolide (MK-8109, EC145) for the Treatment of Recurrent or Refractory Solid Tumors (MK-8109-006, EC-FV-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8109-006; EC-FV-01 (Other: Endocyte)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Cancer
Keywords: Cancer; Phase I; EC145; Recurrent; Refractory; Solid Tumors; Experimental
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Vintafolide 1.2 mg IV Bolus (Experimental): Vintafolide 1.2 mg administered by IV bolus on Days 1, 3, 5, 15, 17, and 19 of 4-week treatment cycles
  Interventions: Drug: Vintafolide IV Bolus
- Vintafolide 2.5 mg IV Bolus (Experimental): Vintafolide 2.5 mg administered by IV bolus on Days 1, 3, 5, 15, 17, and 19 of 4-week treatment cycles
  Interventions: Drug: Vintafolide IV Bolus
- Vintafolide 4.0 mg IV Bolus (Experimental): Vintafolide 4.0 mg administered by IV bolus on Days 1, 3, 5, 15, 17, and 19 of 4-week treatment cycles
  Interventions: Drug: Vintafolide IV Bolus
- Vintafolide 2.5 mg IV Infusion (Experimental): Vintafolide 2.5 mg administered by a 1-hour IV infusion on Days 1, 3, 5, 15, 17, and 19 of 4-week treatment cycles
  Interventions: Drug: Vintafolide IV Infusion
- Vintafolide 3.0 mg IV Infusion (Experimental): Vintafolide 3.0 mg administered by a 1-hour IV infusion on Days 1, 3, 5, 15, 17, and 19 of 4-week treatment cycles
  Interventions: Drug: Vintafolide IV Infusion

INTERVENTIONS:
Drug: Vintafolide IV Bolus — Vintafolide is a folic acid desacetylvinblastine hydrazide conjugate
  Arms: Vintafolide 1.2 mg IV Bolus; Vintafolide 2.5 mg IV Bolus; Vintafolide 4.0 mg IV Bolus
Drug: Vintafolide IV Infusion — Vintafolide is a folic acid desacetylvinblastine hydrazide conjugate
  Arms: Vintafolide 2.5 mg IV Infusion; Vintafolide 3.0 mg IV Infusion

SUMMARY:
This is a Phase I clinical trial evaluating the safety and tolerability of escalating doses of vintafolide (EC145) in participants with relapsed or refractory advanced tumors. The primary objective of this study is to determine the safety and maximum tolerated dose of vintafolide given by intravenous bolus or infusion. The efficacy of the treatment will also be measured.

DETAILED DESCRIPTION:
This is a dose escalation study of vintafolide administered by intravenous (IV) bolus or infusion during weeks 1 and 3 of a 4-week cycle to participants with solid tumors refractory to current therapies. Vintafolide is a drug that is specifically designed to enter cells via a folate vitamin receptor. Experimental evidence shows that the target receptor is over-expressed in many human cancers. There are no previous human studies of vintafolide treatment; however, lab research (research in test tubes and/or animals) using vintafolide has shown activity against tumors in animals. This activity in animal models suggests that vintafolide may be useful as chemotherapy against human cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of neoplasm
* No effective standard therapeutic options
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* >=4 weeks post therapeutic radiation of chemotherapy >=6 weeks for nitrosoureas and mitomycin C) and recovery from associated toxicities
* Negative serum pregnancy test for women of child-bearing potential and willingness to practice contraceptive methods
* Adequate bone marrow reserve, renal, and hepatic function

Exclusion Criteria:

* Concurrent hematological malignancies
* Women who are pregnant or lactating
* Evidence of symptomatic brain metastases
* Receiving concomitant anticancer therapy (excluding supportive care)
* Requires palliative radiotherapy at time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose During Cycle 1 Treatment | Up to Day 26 in Treatment Cycle 1
  Maximum Tolerated Dose (MTD) was defined as the highest dose that can safely be administered to a patient to produce acceptable, manageable and reversible toxicity. This level was further defined as the dose level at which no more than 1 of 6 participants had dose-limiting toxicity (DLT) and the level below the dose at which ≥2 of 6 participants had DLT.

SECONDARY OUTCOMES:
Number of Participants with Best Overall Tumor Response: Participants with Folate Receptor Positive Tumors at Baseline | Up to Week 24
  Tumor status was assessed according to Response Evaluation Criteria in Solid Tumors. Tumor responses used as a reference the sum of the longest diameter (LD) of the target lesions using imaging studies. Partial Response was defined as ≥30% decrease in LD. Stable Disease was defined as neither sufficient shrinkage or increase in LD to qualify as either Partial Response or Progressive Disease. Progressive Disease was defined as ≥20% increase in LD.
Number of Participants with a Dose-Limiting Toxiciity During Cycle 1 Treatment | Up to Day 26 in Treatment Cycle 1
  Dose limiting toxicity was defined as an adverse event that is likely related to the study medication, and fulfills any one of the following criteria: Grade 2 non-hematological toxicity that fails to recover to a Grade 1 level or Baseline at the time that the next treatment cycle is due (with the exception of alopecia); Grade 3 non-hematological toxicity (except for nausea/vomiting without maximal symptomatic / prophylactic treatment); Grade 4 hematological toxicity; Toxicity that, in the opinion of the investigator, would prevent use of the drug dose or regimen by the general oncology community.
Number of Participants with an Adverse Event Leading to Study Discontinuation During Cycle 1 Treatment | Up to Day 26 in Treatment Cycle 1
  An adverse event was defined as any untoward, undesired, or unplanned clinical event in the form of physical signs, symptoms, disease, laboratory or physiological observations in a participant administered the Sponsor's product whether or not related to the use of the product
Number of Participants with Best Overall Tumor Response: All Treated Participants | Up to Week 24
  Tumor status was assessed according to Response Evaluation Criteria in Solid Tumors. Tumor responses used as a reference the sum of the longest diameter (LD) of the target lesions using imaging studies. Complete Response was defined as disappearance of all target lesions. Partial Response was defined as ≥30% decrease in LD. Stable Disease was defined as neither sufficient shrinkage or increase in LD to qualify as either Partial Response or Progressive Disease. Progressive Disease was defined as ≥20% increase in LD.
Maximum Plasma Concentration (Cmax) of Vintafolide on Day 1 of Treatment Cycle 1 | Up to 90 minutes after IV bolus dosing and up to 60 minutes after the start of the 1-hour IV infusion on Day 1 of treatment cycle 1
  Blood was collected from participants for determination of plasma vintafolide. The lower limit of quantitation for vintafolide was 10 ng/mL.
Maximum Plasma Concentration (Cmax) of Vintafolide on Day 3 of Treatment Cycle 1 | Up to 90 minutes after IV bolus dosing and up to 60 minutes after the start of the 1-hour IV infusion on Day 3 of treatment cycle 1
  Blood was collected from participants for determination of plasma vintafolide. The lower limit of quantitation for vintafolide was 10 ng/mL.
Area Under the Plasma Concentration-Time Curve (AUC) of Vintafolide on Day 1 of Treatment Cycle 1 | Up to 90 minutes after IV bolus dosing and up to 60 minutes after the start of the 1-hour IV infusion on Day 1 of treatment cycle 1
  Blood was collected from participants for determination of plasma vintafolide. The lower limit of quantitation for vintafolide was 10 ng/mL.
Area Under the Plasma Concentration-Time Curve (AUC) of Vintafolide on Day 3 of Treatment Cycle 1 | Up to 90 minutes after IV bolus dosing and up to 60 minutes after the start of the 1-hour IV infusion on Day 3 of treatment cycle 1
  Blood was collected from participants for determination of plasma vintafolide. The lower limit of quantitation for vintafolide was 10 ng/mL.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- [Result] Li J, Sausville EA, Klein PJ, Morgenstern D, Leamon CP, Messmann RA, LoRusso P. Clinical pharmacokinetics and exposure-toxicity relationship of a folate-Vinca alkaloid conjugate EC145 in cancer patients. J Clin Pharmacol. 2009 Dec;49(12):1467-76. doi: 10.1177/0091270009339740. Epub 2009 Oct 16. PMID 19837906
- [Result] Lorusso PM, Edelman MJ, Bever SL, Forman KM, Pilat M, Quinn MF, Li J, Heath EI, Malburg LM, Klein PJ, Leamon CP, Messmann RA, Sausville EA. Phase I study of folate conjugate EC145 (Vintafolide) in patients with refractory solid tumors. J Clin Oncol. 2012 Nov 10;30(32):4011-6. doi: 10.1200/JCO.2011.41.4946. Epub 2012 Oct 1. PMID 23032618